CLINICAL TRIAL: NCT04551885
Title: A Phase I, Open-Label, Multicenter Study of FT516 in Combination With Monoclonal Antibodies in Subjects With Advanced Solid Tumors
Brief Title: FT516 in Combination With Monoclonal Antibodies in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated by the Sponsor.
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT516-102
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor, Adult
Keywords: PD-L1; cellular therapy; NK cells; urothelial cancer; renal cell carcinoma; merkel cell carcinoma; non-small cell lung cancer; NSCLC; triple negative breast cancer; immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Merkel Cell; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms | interventions — avelumab; Cyclophosphamide; fludarabine; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FT516 in combination with avelumab (Experimental)
  Interventions: Drug: FT516; Drug: Avelumab; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2

INTERVENTIONS:
Drug: FT516 — Experimental Interventional Therapy
Drug: Avelumab — Monoclonal antibody
  Other Names: Bavencio
Drug: Cyclophosphamide — Lympho-conditioning agent
Drug: Fludarabine — Lympho-conditioning agent
Drug: IL-2 — Biologic response modifier
  Other Names: Proleukin; Aldesleukin

SUMMARY:
This is a Phase 1 dose-finding study of FT-516 in combination with monoclonal antibodies in participants with advanced solid tumors. The study will consist of a dose-escalation stage and an expansion stage where participants will be enrolled into indication-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic solid tumor malignancies that have relapsed or progressed after at least one line of therapy and where the following anti-PD-L1 are approved: avelumab, atezolizumab or durvalumab
* Capable of giving signed informed consent
* Aged ≥ 18 years old
* Willingness to comply with study procedures and duration
* Measurable disease per iRECIST
* Contraceptive use for women and men as defined in the protocol

Exclusion Criteria:

* Pregnant or breast-feeding women
* ECOG performance status ≥ 2
* Evidence of insufficient organ function
* Clinically significant cardiovascular disease
* Receipt of therapy within 2 weeks prior to Day 1 or five half-lives, whichever is shorter or any investigational therapy within 28 days prior to Day 1
* Known active central nervous system (CNS) involvement by malignancy
* Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis or neurodegenerative disease or receipt of medications for these conditions
* Currently receiving or likely to require immunosuppressive therapy
* Known active infections with Hepatitis B, Hepatitis C or HIV
* Live vaccine within 6 weeks prior to start of lympho-conditioning
* Known allergy to albumin (human) or DMSO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) Within Each Dose Level Cohort | Up to Day 29 after the end of Cycle 1 (each cycle is 28 days)
  The incidence of DLTs within each dose level cohort will be reported. A DLT is any adverse event (AE) that is at least possibly related to FT516 that occurs after the first FT516 infusion through the end of the DLT assessment period on Cycle 1 Day 29, and meets 1 of the criteria from the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 or the American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading Guidelines for Cytokine Release Syndrome and Neurological Toxicity Associated with Immune Effector Cells.
Severity of DLTs Within Each Dose Level Cohort | At the end of Cycle 1 (each cycle is 28 days)
  The severity of DLTs within each cohort will be reported. DLT is any adverse event (AE) that is at least possibly related to FT516 that occurs after the first FT516 infusion through the end of the DLT assessment period on Cycle 1 Day 29, and meets 1 of the criteria from the NCI CTCAE v5.0 or the ASTCT Consensus Grading Guidelines for Cytokine Release Syndrome and Neurological Toxicity Associated with Immune Effector Cells.

SECONDARY OUTCOMES:
Number of Participants with ≥1 Adverse Events (AE) | Up to 15 years
  An AE is any untoward medical occurrence in a participants temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Investigator-Assessed Duration of Response (DOR) | Up to 15 years
  DOR is the time from the first occurrence of a documented, objective response until the time of disease progression, relapse or death from any cause, whichever occurs first, per modified Response Evaluation Criteria in Solid Tumors (iRECIST) response criteria.
Disease Control Rate (DCR) | Up to 15 years
  DCR is defined as the percentage of participants with Stable Disease more than 6 months, Partial Response or Complete Response, per iRECIST response criteria.
Progression Free Survival (PFS) | Up to 15 years
  PFS is defined as the time from first dose of lympho-conditioning to disease progression or to the day of death for any reason, whichever occurs first, per iRECIST response criteria.
Overall Survival (OS) | Up to 15 years
  OS is defined as the time from first dose of lympho-conditioning to death from any cause.
Determination of PK of FT516 in peripheral blood | Study Days 1, 2, 4, 8, 11, 18, 22, 29
  The pharmacokinetics of FT516 in peripheral blood will be reported as the relative percentage of product (FT516) DNA versus patient DNA (% chimerism) measured from blood samples at the specified time points

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics
Locations (3):
- United States (3):
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Hackensack University Medical Center/John Theurer Cancer Center, Hackensack, New Jersey
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu H, Blum RH, Bjordahl R, Gaidarova S, Rogers P, Lee TT, Abujarour R, Bonello GB, Wu J, Tsai PF, Miller JS, Walcheck B, Valamehr B, Kaufman DS. Pluripotent stem cell-derived NK cells with high-affinity noncleavable CD16a mediate improved antitumor activity. Blood. 2020 Feb 6;135(6):399-410. doi: 10.1182/blood.2019000621. PMID 31856277